CLINICAL TRIAL: NCT06177587
Title: Multimarker Evaluation of Platelet Activity and Agregation in Patients Presenting With Acute Coronary Syndrome: Prospective Observational Study
Brief Title: Multimarker Evaluation of Platelet Activity and Agregation in ACS
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Mariusz Tomaniak, Tomaniak Mariusz MD PhD, Medical University of Warsaw
Other Study IDs: MULTIMARKER-ACS
Record Dates: First submitted 2023-12-08; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Syndrome; Biomarkers; IPF; Immature Platelet Fraction; ADP test; Antiplatelet therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Assesment of platelet biomarkers in acute coronary syndromes - low level of parameters: Blood is collected within the first 24 hours from hospital admission and after 72 hours following hospital admission. The level of selected biomarkers is measured.
  Interventions: Other: Assesment of biomarkers in acute coronary syndromes
- Assesment of platelet biomarkers in acute coronary syndromes - high level of parameters: Blood is collected within the first 24 hours from hospital admission and after 72 hours following hospital admission. The level of selected biomarkers is measured.
  Interventions: Other: Assesment of biomarkers in acute coronary syndromes

INTERVENTIONS:
Other: Assesment of biomarkers in acute coronary syndromes — Collection of 20ml of blood from peripheral vein.

SUMMARY:
Patients with acute coronary syndrome (ACS) who undergo percutaneous coronary intervention (PCI) are at a higher risk of ischemic complications, even while receiving proper dual antiplatelet therapy. For this reason, identifying high-risk patients and personalizing treatment according to their profile could be a solution towards improving the efficacy and safety of the antiplatelet treatment.

This is a prospective single centre study analyzing correlations and clinical outcomes of patients in relation to biomarkers in acute coronary syndrome. The blood samples were collected from patients admitted to the hospital with a diagnosis of ACS and treated with dual antiplatelet therapy.

The blood samples were collected from each patient within the first 24 hours after the admission for acute coronary syndrome (ACS) and after 72 hours of hospitalization.

DETAILED DESCRIPTION:
In this prospective, single-center, observational study, adult patients meeting the inclusion/exclusion criteria were included. Subjects enrolled at the Invasive Cardiology Unit of the 1st Department of Cardiology; Medical University of Warsaw (Poland) were cathegorized into three arms: 1) treated with aspirin and clopidogrel, 2) treated with aspirin and ticagrelor; 3) treated with aspirin and prasugrel. In all three groups subjects first obtained the loading dose of the drug and thereafter they received a fixed daily dose.

Blood samples were collected form each patient at two time-points: during the first 24 hours from hospital admission and after 72 hours following hospital admission. The parameters measured included selected platelet-derived microRNAs prticles, immature platelet fraction (IPF) and platelet microvesicles' comncentration. Platelet reactivity was established using Multiplate® Analyzer (Roche).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent in a time window 1-24 hours after successful PCI;
2. Male or female, age ≥ 18 years at screening;
3. ACS at the time of the index hospitalization;
4. ACS patients undergoing PCI (New-Generation DES)
5. Use of a loading dose of P2Y12 inhibitor administered after diagnosis of ACS or after PCI;

Exclusion Criteria:

1. Unstable clinical status (hemodynamic or electrical instability);
2. Planned surgery requiring DAPT discontinuation during the study;
3. Coronary Revascularization (Surgical or Intervention) Program within 90 days
4. Prior stroke, transient ischemic attack or intracranial bleeding;
5. Active bleeding;
6. Severe anemia (hemoglobin < 8g/dL);
7. Platelet count ≤70x10^3/ml;
8. Hematocrit of < 30% or > 52%
9. Renal failure (hemodialysis or creatinine clearance ≤ 30 ml/min calculated with Cockroft-Gault formula);
10. Severe hepatic dysfunction (baseline alanine aminotransferase ≥ 2.5 times the upper limit of normal);
11. Known hypersensitivity or contraindication to ASA, clopidogrel, ticagrelor or prasugrel;
12. Under judicial protection, tutorship or curatorship;
13. Pregnancy;
14. Unable to understand and follow study-related instructions;
15. Enrollment in another investigational device or drug study.
16. Unable to provide an informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population diagnosed with ACS on admission and treated primarily with PCI.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Correlation between the selected biomarkers in patients with acute coronary syndrome in the first 24 hours from hospital admission and major adverse cardiovascular events (MACE) | 50 months
  MACE defined as the composite endpoint of all-cause death, myocardial infarction, stroke, unplanned revascularization.

CONTACTS AND LOCATIONS:
Locations (1):
- I Department and Clinic of Cardiology, Medical University of Warsaw, Warsaw, Poland

REFERENCES:
- [Derived] Gumiezna K, Bednarek A, Sygitowicz G, Maciejak-Jastrzebska A, Barus P, Hunia J, Klimczak-Tomaniak D, Kochman J, Grabowski M, Tomaniak M. Platelet microRNAs as Potential Novel Biomarkers for Antiplatelet Therapy with P2Y12 Inhibitors and Their Association with Platelet Function. J Clin Med. 2023 Dec 22;13(1):63. doi: 10.3390/jcm13010063. PMID 38202070
- [Derived] Gumiezna K, Barus P, Sygitowicz G, Wisniewska A, Bednarek A, Zablocki J, Piasecki A, Klimczak-Tomaniak D, Kochman J, Grabowski M, Tomaniak M. Prognostic Implications of Immature Platelet Fraction at 5-Year Follow-up Among ACS Patients Treated With Dual Antiplatelet Therapy. J Cardiovasc Pharmacol Ther. 2024 Jan-Dec;29:10742484231202864. doi: 10.1177/10742484231202864. PMID 38196286
- [Derived] Gumiezna K, Bednarek A, Sygitowicz G, Barus P, Wisniewska A, Klimczak-Tomaniak D, Kochman J, Opolski G, Grabowski M, Tomaniak M. Immature platelet fraction and immature platelet count as novel biomarkers of elevated platelet reactivity in NSTE-ACS patients receiving dual antiplatelet therapy. Adv Clin Exp Med. 2023 Dec;32(12):1465-1470. doi: 10.17219/acem/177406. PMID 38126718